CLINICAL TRIAL: NCT06270524
Title: Pilot Study of the C5a/C5aR1 Axis in IgG4-associated Disease: a Potential Therapeutic Target. C5-MAG4 Study.
Brief Title: Study of the C5a/C5aR1 Axis in IgG4-associated Disease: a Potential Therapeutic Target
Acronym: C5-MAG4
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RCAPHM21_0433
Record Dates: First submitted 2024-02-14; First posted 2024-02-21 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Immunoglobulin G4-Related Disease
MeSH Terms: conditions — Immunoglobulin G4-Related Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IgG4-RD patient (Experimental): Patients suffering from Immunoglobulin G4-related disease (IgG4-RD).
  Interventions: Procedure: Blood sampling
- patient in remission (Experimental): Patients suffering from Immunoglobulin G4-related disease (IgG4-RD) but in remission.
  Interventions: Procedure: Blood sampling
- healthy volunteers (Other)
  Interventions: Procedure: Blood sampling

INTERVENTIONS:
Procedure: Blood sampling — Blood sampling will be taken for further analysis

SUMMARY:
This is a monocentric, comparative, cross-sectional, case-control study seeking to identify abnormalities of the C5a-C5aR1 axis between a population of patients with active IgG4-associated disease (MAG4) and two control groups: healthy subjects without MAG4 and patients with MAG4 in remission.

DETAILED DESCRIPTION:
IgG4-associated disease is a rare fibrosing and inflammatory disorder whose pathophysiology remains poorly understood. Activation of certain monocyte/macrophage populations (in particular M2-type macrophages) has been shown to be involved during the course of the disease. The mechanisms behind this monocyte/macrophage activation are not known. Expression of the C5aR receptor on the surface of these populations, and preliminary findings of elevated C5a in these patients, suggest a potential role for this C5a-C5aR axis. Demonstration of the involvement of this pathway would open a path to therapeutic perspetives (C5aR inhibitors) for these patients, who frequently suffer from cortico-dependence and relapses. The aim of this research is to use healthcare technologies to identify cellular and molecular therapeutic targets in the context of the IgG4-associated disease

ELIGIBILITY:
Inclusion Criteria for patients suffering from IG4-related disease and patients in remission :

* age > 18
* diagnosis of IgG4-associated disease according to ACR/EULAR 2019 classification criteria (4,5) with a score ≥20.
* disease activity score (IgG4-RD Responder Index) ≥2 in at least one affected organ

Exclusion Criteria for patients suffering from IG4-related disease and patients in remission :

* presence of a differential diagnosis ("IgG4-RD mimicker") or exclusion criterion according to ACR/EULAR 2019 classification criteria (4,5).
* systemic corticosteroid treatment ≥5 mg/day ongoing or < 1 month ; Study C5-MAG4_RCAPHM21_0433 Protocol Version 1.1 of 16/01/2024 Page 15 of 41
* immunosuppressive therapy ongoing or < 3 months ;
* current biotherapy treatment or < 6 months;
* absence of signed informed consent;
* absence of affiliation to a Social Security scheme.
* patient participating in an ongoing therapeutic trial ;
* any condition which, in the opinion of the investigator, could influence the results of the study.

Inclusion criteria for healthy volunteers :

- age > 18

Exclusion criteria for healthy volunteers :

* infectious episode (temperature >38°C, flu-like signs) in the 30 days prior to inclusion;
* known inflammatory (including IG4-related disease) or autoimmune pathology;
* treatment with corticosteroids in progress or taken in the month prior to sampling, or immunosuppressants in progress or taken in the 3 months prior to sampling, or biotherapy in the 6 months prior to sampling;
* absence of signed informed consent;
* absence of affiliation to a Social Security scheme;
* persons taking part in an ongoing therapeutic trial;
* any condition which, in the opinion of the investigator, could influence the results of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Serum C5a concentration | 24 months
  The C5a concentration in the serum will be compared between of healthy volunteers and patients suffering from IG4-related disease

SECONDARY OUTCOMES:
frequency of C5aR1+ monocytes among total monocytes | 24 months
  The frequency of C5aR1+ monocytes among total monocytes will be compared between :
  * patients suffering from IG4-related disease and healthy volunteers
  * patients suffering from IG4-related disease and patients in remission
frequency of Tumor Growth Factor B+ (TGF-B+) monocytes among total monocytes | 24 months
  frequency of Tumor Growth Factor B+ (TGF-B+) monocytes among total monocytesill be compared between :
  * patients suffering from IG4-related disease and healthy volunteers
  * patients suffering from IG4-related disease and patients in remission